CLINICAL TRIAL: NCT05999461
Title: Association of Auditory Dysfunction With Retinal Ischemia in Behcet Disease
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maha Sayed Ibrahim Abdelrahman, Principal investigator, Assiut University
Other Study IDs: behcet disease
Record Dates: First submitted 2023-08-12; First posted 2023-08-21 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Behcet's Disease With Multisystem Involvement

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases: behcet patients
- control: age and sex matched healthy volunteers

SUMMARY:
Auditory dysfunction is commonly detected in Behçet's disease (BD). Also, vestibular abnormalities as well as cochlear function affection have been found. The inflammatory process in BD may be the cause of audiometry abnormalities in those patients. The aim of this study is to assess hearing dysfunction in Behçet patients and its relation to retinal ischemia and disease activity using conventional pure-tone audiometry (cPTA), tympanogram and acoustic reflex

DETAILED DESCRIPTION:
pure tone audiometry is a behavioral test used to measure hearing sensitivity. This measure involves the peripheral and central auditory systems. Pure-tone thresholds (PTTs) indicate the softest sound audible to an individual at least 50% of the time. Hearing sensitivity is plotted on an audiogram, which displays intensity as a function of frequency.

Speech audiometry employs speech signals to assess if the patient has problems hearing speech or speech in noise. Speech audiometry can be used to examine the processing ability and if it is affected by disorders of the middle ear, cochlea, auditory nerve, brainstem pathway, or auditory centers of the cortex.

Tympanogram is a test of middle ear functioning. This objective test also allows to view the functioning of the Eustachian Tube, the upper auditory pathways and the reflex contraction from the middle ear muscles. Impedance testing is crucial in distinguishing a conductive loss from a sensorineural hearing loss.

Optical coherence tomography angiography (OCT-A) for imaging the microvasculature of the retina and the choroid.

Behcet disease current activity form for assessment of disease activity range from 0 to 12 . 12 represents the highest disease activity. It depends on the symptoms present over the last 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* All patients fulfill the International Criteria of behcet disease

Exclusion Criteria:

* age more than 50
* ear infection,
* ear trauma, acoustic trauma, or usage of ototoxic drugs.
* Also, associated systemic diseases that can affect the hearing as infectious diseases (e.g., mumps, CMV), granulomatous diseases (e.g., sarcoidosis, Wegner's granulomatosis), other autoimmune diseases (e.g., Rheumatoid arthritis, Cogan's syndrome, polyarteritis nodosa, relapsing polychondritis), and diseases of the bone (e.g., Paget's disease).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study subjects consist of 2 groups. the first group is behcet patients that fulfill the International Criteria of behcet disease. second group consists of age and sex matched healthy volunteers
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Detection of hearing abnormalities in behcet disease | 3 MONTHS
  pure tone audiometry, tympanogram and acoustic reflex
correlation of hearing abnormalities with retinal ischemia | 3 months
  oct angiography

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt